CLINICAL TRIAL: NCT06723912
Title: The Effect of Health Action Process Approach-Based Program on Hemodialysis Patients' Adherence to Treatment and Quality of Life
Brief Title: Implementation of a Health Action Process Approach-Based Program for People on Hemodialysis Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Yelda KOÇAK, PhD student, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: YKOCAK
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-11

CONDITIONS: Hemodialytic Patients
Keywords: Health action process approach; hemodialysis; quality of life; treatment adherence; care
MeSH Terms: conditions — Treatment Adherence and Compliance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (No Intervention): No program will be applied to the control group. Routine treatment and care in the hospital will continue. At the end of the study, a Handbook for Adherence to Hemodialysis Treatment will be given.
- Intervention Group (Experimental): Program based on the Health Action Process Approach will be implemented. Hemodialysis Treatment Compliance Handbook will be given.
  Interventions: Other: Health Action Process Approach-Based Program

INTERVENTIONS:
Other: Health Action Process Approach-Based Program — Health Action Process Approach-Based Program: The program is planned for six weeks (six sessions). Sessions will be held once a week for 30-45 minutes. Within the scope of the program, care - structured nursing care plans based on the Health Action Process Approach will be made -, education and counseling will be provided. Sessions will be held in a quiet, calm environment in the hospital, and if such an environment cannot be provided, they will be held at the patient's home. The day, time and place of the sessions will be decided together with the participant after each interview or session. At the beginning of each session, the previous session will be briefly recalled and the homework (SWOT analysis, treatment adherence tracking chart or SMART goal plan) given in the previous session will be evaluated. At the end of each session, the evaluation of that day's session will be carried out briefly.
  Arms: Intervention Group

SUMMARY:
The aim of the study is to determine the effect of the Health Action Process Approach (HAPA) based program on the treatment compliance and quality of life of people undergoing hemodialysis treatment. The hypotheses of the study are as follows:

* The Health Action Process Approach Based Program has an effect on the treatment compliance of people undergoing hemodialysis treatment.
* The Health Action Process Approach Based Program has an effect on the quality of life of people undergoing hemodialysis treatment.
* The Health Action Process Approach Based Program has an impact on the results of laboratory tests and clinical parameters of people receiving hemodialysis treatment.

The population of the study will consist of people receiving hemodialysis treatment in the main service building and additional service building of Kahramanmaraş Necip Fazıl City Hospital. Patients who meet the criteria of ''volunteering to participate in the study, being over the age of 18, being literate, not having any problems that may prevent communication, not having a history of neurological or psychiatric disease, being on hemodialysis treatment for at least six months, and the vascular access used for hemodialysis being effective'' will be included in the study. Written informed consent will be obtained from patients who volunteer to participate in the study. At least 32 people who meet the inclusion criteria will be included in each group. The intervention group will receive a program based on the Health Action Process Approach (HAPA). No program will be applied to the control group.

The data collection tools of the study consist of the Participant Information Form, Participant Evaluation Form Based on the Health Action Process Approach, End-Stage Renal Disease Adherence Scale (ESRD-AQ), Fluid Control Scale in Hemodialysis Patients, Diet Information Scale of Hemodialysis Patients, Diet Behavior Scale of Hemodialysis Patients, Quality of Life (SF-36) Form, Laboratory Tests Follow-up Form and Homework Form. Measurements of the groups will be taken at the beginning of the study, week 6 (at the end of the program), month 3 and month 6.

DETAILED DESCRIPTION:
The Health Action Process Approach (HAPA) Model was developed by Ralf Schwarzer in 1992 to understand the process of health behavior change. The Health Action Process Approach Model focuses on the "intention-behavior gap", which states that intentions to perform the behavior are sometimes not sufficient to take action to perform the behavior. Other social cognitive models are criticized for this "intention-behavior gap". Because in most of these models, it is stated that intention is the most important predictor for behavior change, and if the intention to perform the behavior is formed, the behavior will occur; however, intentions do not always turn into behavior. In order to close the intention-behavior gap, the HAPA Model proposes to evaluate the pre-intention motivation processes that lead to behavioral intention and the post-intention volitional processes that lead to behavior in two separate stages. The motivation stage of the model includes the components of "risk perception", "outcome expectations" and "action self-efficacy" and it is thought that the formation of behavioral intention depends on these components. The volitional stage of the model includes "action planning", "coping planning", "coping self-efficacy", "improvement self-efficacy" and "social support" and these are effective in the realization and maintenance of health behaviors. The HAPA Model is an important model in terms of providing a detailed and comprehensive description of the motivation processes before the formation of health behavior intention, the transformation of intention into behavior and the maintenance of behavior within these components. The volitional stage of the model includes "action planning", "coping planning", "coping self-efficacy", "improvement self-efficacy" and "social support" and these are effective in the realization and maintenance of health behaviors. The HAPA Model is an important model in terms of providing a detailed and comprehensive description of the motivation processes before the formation of health behavior intention, the transformation of intention into behavior and the maintenance of behavior within these components.

Health Action Process Approach-Based Program: The program is planned for six weeks (six sessions). Sessions will be held once a week for 30-45 minutes. Within the scope of the program, care - structured nursing care plans based on the Health Action Process Approach will be made -, education and counseling will be provided. Sessions will be held in a quiet, calm environment in the hospital, and if such an environment cannot be provided, they will be held at the patient's home. The day, time and place of the sessions will be decided together with the participant after each interview or session. At the beginning of each session, the previous session will be briefly recalled and the homework (SWOT analysis, treatment adherence tracking chart or SMART goal plan) given in the previous session will be evaluated. At the end of each session, the evaluation of that day's session will be carried out briefly.

In the study, two groups will be formed as intervention and control groups. No program will be applied to the intervention group. Routine treatment and care will continue. The control group will receive routine treatment and care as well as a program based on the Health Action Process Approach. Hemodialysis Treatment Adherence Handbook will be given to the intervention group when the study is completed. Participants in both groups will fill out the Health Action Process Approach-Based Participant Evaluation Form, Laboratory Tests Monitoring Form, End Stage Renal Failure Compliance Scale, Fluid Control Scale in Hemodialysis Patients, Dietary Knowledge Scale of Hemodialysis Patients, Dietary Behavior Scale of Hemodialysis Patients and Quality of Life (SF-36) Form. These forms will be completed at the beginning of the study (week 0), week 6 (at the end of the program), month 3 and month 6.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Over 18 years of age
* Being literate
* Not having any problems with speech, hearing or vision that may interfere with communication
* No history of neurological or psychiatric disease
* Being on hemodialysis treatment for at least six months
* The vascular access (catheter, fistula or graft) used to administer hemodialysis is working effectively

Exclusion Criteria:

* Not meeting the inclusion criteria
* Participation in a program based on the Health Action Process Approach related to the subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-10-23 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Changes in the attendance of people receiving hemodialysis treatment at hemodialysis sessions | Beginning of the study (week 0), week 6 (at the end of the program), 3rd month, and 6th month
  Health Action Process Approach Based Participant Evaluation Form: It is a form created by the researcher based on the studies in the literature. There are 11 questions regarding participation in hemodialysis sessions. The questions can be answered "yes", "partially" and "no".
Changes in adherence to dietary restriction in people receiving hemodialysis treatment | Beginning of the study (week 0), week 6 (at the end of the program), 3rd month, and 6th month
  Health Action Process Approach Based Participant Evaluation Form: It is a form created by the researcher based on the studies in the literature. There are 11 questions regarding the compliance of people receiving hemodialysis treatment with dietary restriction. The questions can be answered "yes", "partially" and "no".
Changes in compliance with fluid restriction in people on hemodialysis | Beginning of the study (week 0), week 6 (at the end of the program), 3rd month, and 6th month
  Health Action Process Approach Based Participant Evaluation Form: It is a form created by the researcher based on the studies in the literature. There are 11 questions regarding the compliance of people receiving hemodialysis treatment with fluid restriction. The questions can be answered "yes", "partially" and "no".
Changes in adherence to medication use among people receiving hemodialysis treatment | Beginning of the study (week 0), week 6 (at the end of the program), 3rd month, and 6th month
  Health Action Process Approach Based Participant Evaluation Form: It is a form created by the researcher based on the studies in the literature. There are 11 questions regarding the medication compliance of people receiving hemodialysis treatment. The questions can be answered "yes", "partially" and "no".
Change in adherence of people on hemodialysis treatment | Beginning of the study (week 0), week 6 (at the end of the program), 3rd month, and 6th month
  End-Stage Renal Disease Adherence Questionnaire (ESRD-AQ): The scale consists of four sections: participation in haemodialysis treatment, medication use, fluid restriction and dietary restriction. A score between 0-1200 can be obtained from the scale. The increase in the score obtained from the scale indicates an increase in treatment compliance. There are no reverse coded items in the scale. Since the items in the scale do not have a homogenous structure, Cronbach's alpha coefficient cannot be calculated.
Change in treatment adherence (dietary adherence) of people receiving hemodialysis treatment | Beginning of the study (week 0), week 6 (at the end of the program), 3rd month, and 6th month
  Dietary Knowledge Scale of Hemodialysis Patients: It was used to evaluate the dietary compliance of people undergoing haemodialysis treatment in detail. The scale has a 3-point Likert type. The questions can be answered as ''true'', ''false'' and ''don't know''. The answers are scored as 1, 0 and 0 respectively. There are no reverse coded items. Scores between 0-18 can be obtained from the scale. The increase in the score indicates that the level of knowledge is good. Cronbach Alpha value is 0.86.
Change in treatment adherence (dietary adherence) of people receiving hemodialysis treatment | Beginning of the study (week 0), week 6 (at the end of the program), 3rd month, and 6th month
  Dietary Behaviour Scale of Hemodialysis Patients: It was used to evaluate the dietary compliance of people undergoing haemodialysis treatment in detail. The scale consists of one sub-dimension and 13 items. The items are scored as ''strongly disagree=1, disagree= 2, undecided= 3, agree= 4, strongly agree= 5''. There are no items that need to be reverse coded. A score between 13-65 can be obtained from the scale. A high score indicates that the behavioural status is 'good'.
Change in adherence to treatment (adherence to fluid restriction) of people receiving hemodialysis treatment | Beginning of the study (week 0), week 6 (at the end of the program), 3rd month, and 6th month
  Fluid Control Scale in Haemodialysis Patients: It was used to evaluate in detail the compliance of people on haemodialysis treatment with fluid restriction. The scale consists of 24 items and three sub-dimensions (knowledge-behaviour-attitude). The items are scored as ''agree=3, undecided=2, disagree=1''. Items 6, 7, 18, 19, 20, 21, 22, 23, 24 are scored by reverse coding. A score between 24-72 can be obtained from the scale. The increase in the score obtained from the scale indicates that the fluid control of the patients also increases.
Change in the quality of life of people undergoing hemodialysis treatment | Beginning of the study (week 0), week 6 (at the end of the program), 3rd month, and 6th month
  Quality of Life (SF-36) Form: It was used to assess the quality of life of people undergoing haemodialysis treatment. The scale consists of eight sub-dimensions (physical function, social function, pain, vitality (energy), role limitation-emotional, role limitation-physical, mental health, general perception of health) and 36 items. The total score of the scale is not calculated and the total scores of the sub-dimensions are calculated separately. The scores that can be obtained vary between 0-100. A high score indicates a high quality of life.
Change in URR value of people on haemodialysis treatment | Beginning of the study (week 0), week 6 (at the end of the program), 3rd month, and 6th month
  It will be taken from the patient file.
Change in haemoglobin value of people undergoing haemodialysis treatment | Beginning of the study (week 0), week 6 (at the end of the program), 3rd month, and 6th month
  It will be taken from the patient file.
Change in potassium value of people undergoing haemodialysis treatment | Beginning of the study (week 0), week 6 (at the end of the program), 3rd month, and 6th month
  It will be taken from the patient file.
Change in sodium value of people undergoing haemodialysis treatment | Beginning of the study (week 0), week 6 (at the end of the program), 3rd month, and 6th month
  It will be taken from the patient file.
Change in creatinine value of people on haemodialysis treatment | Beginning of the study (week 0), week 6 (at the end of the program), 3rd month, and 6th month
  It will be taken from the patient file.
Change in Kt/V value of people receiving haemodialysis treatment | Beginning of the study (week 0), week 6 (at the end of the program), 3rd month, and 6th month
  It will be taken from the patient file.
Change in urea value of people undergoing haemodialysis treatment | Beginning of the study (week 0), week 6 (at the end of the program), 3rd month, and 6th month
  It will be taken from the patient file.
Change in calcium value of people undergoing haemodialysis treatment | Beginning of the study (week 0), week 6 (at the end of the program), 3rd month, and 6th month
  It will be taken from the patient file.
Change in phosphorus value of people undergoing haemodialysis treatment | Beginning of the study (week 0), week 6 (at the end of the program), 3rd month, and 6th month
  Taken from patient file.
Change in glucose value of people undergoing haemodialysis treatment | Beginning of the study (week 0), week 6 (at the end of the program), 3rd month, and 6th month
  It will be taken from the patient file.
Change in total protein value of people on haemodialysis treatment | Beginning of the study (week 0), week 6 (at the end of the program), 3rd month, and 6th month
  It will be taken from the patient file.
Change in MCH value of people undergoing haemodialysis treatment | Beginning of the study (week 0), week 6 (at the end of the program), 3rd month, and 6th month
  It will be taken from the patient file.
Changes in ALT values of people undergoing haemodialysis treatment | Beginning of the study (week 0), week 6 (at the end of the program), 3rd month, and 6th month
  It will be taken from the patient file.
Change in RBC value of people undergoing haemodialysis treatment | Beginning of the study (week 0), week 6 (at the end of the program), 3rd month, and 6th month
  It will be taken from the patient file.
Changes in AST values of people undergoing haemodialysis treatment | Beginning of the study (week 0), week 6 (at the end of the program), 3rd month, and 6th month
  It will be taken from the patient file.
Change in albumin value of people undergoing haemodialysis treatment | Beginning of the study (week 0), week 6 (at the end of the program), 3rd month, and 6th month
  It will be taken from the patient file.
Changes in WBC values of people undergoing haemodialysis treatment | Beginning of the study (week 0), week 6 (at the end of the program), 3rd month, and 6th month
  It will be taken from the patient file.
Change in MCV value of people undergoing haemodialysis treatment | Beginning of the study (week 0), week 6 (at the end of the program), 3rd month, and 6th month
  It will be taken from the patient file.
Change in PLT value of people undergoing haemodialysis treatment | Beginning of the study (week 0), week 6 (at the end of the program), 3rd month, and 6th month
  It will be taken from the patient file.
Change in haematocrit value of people undergoing haemodialysis treatment | Beginning of the study (week 0), week 6 (at the end of the program), 3rd month, and 6th month
  It will be taken from the patient file.
Change in blood pressure of a person undergoing hemodialysis treatment | Beginning of the study (week 0), week 6 (at the end of the program), 3rd month, and 6th month
  Blood pressure value at the entrance and exit of hemodialysis will be measured.
Change in the pulse rate of a person receiving hemodialysis treatment | Beginning of the study (week 0), week 6 (at the end of the program), 3rd month, and 6th month
  The person's pulse rate will be measured at the entrance and exit of hemodialysis treatment.
Change in respiratory rate of a person receiving hemodialysis treatment | Beginning of the study (week 0), week 6 (at the end of the program), 3rd month, and 6th month
  The respiratory rate of the person will be measured at the entrance and exit of hemodialysis treatment.
Change in oxygen saturation of a person receiving hemodialysis treatment | Beginning of the study (week 0), week 6 (at the end of the program), 3rd month, and 6th month
  Oxygen saturation will be measured at the entrance and exit of hemodialysis treatment.
Change in body temperature of the person receiving hemodialysis treatment | Beginning of the study (week 0), week 6 (at the end of the program), 3rd month, and 6th month
  Body temperature will be measured at the entrance and exit of hemodialysis treatment.
Change in weight at entry and exit of hemodialysis treatment | Beginning of the study (week 0), week 6 (at the end of the program), 3rd month, and 6th month
  Hemodialysis treatment entry and exit weight will be weighed.
Changes in dry weight of a person undergoing hemodialysis treatment | Beginning of the study (week 0), week 6 (at the end of the program), 3rd month, and 6th month
  The dry weight of the person receiving hemodialysis treatment will be weighed.
Interdialytic weight changes in a person receiving hemodialysis treatment | Beginning of the study (week 0), week 6 (at the end of the program), 3rd month, and 6th month
  The interdialytic weight of the person receiving hemodialysis treatment will be weighed.

CONTACTS AND LOCATIONS:
Locations (1):
- Kahramanmaraş Necip Fazıl City Hospital, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No